CLINICAL TRIAL: NCT02602626
Title: The Acceptability of the HPV Vaccine Postpartum and With Pediatric Well-child Visits: A Pilot Study
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-2178; 5T32HD040672-15 (NIH)
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2015-11

CONDITIONS: Vaccination
Keywords: Human Papillomavirus; HPV; Postpartum

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if women would find it acceptable to receive the HPV vaccine postpartum at the pediatrician's office at the time of their child's two-month well- child visit when offered during the third trimester of pregnancy.

DETAILED DESCRIPTION:
There are a large number of young adult women who have not received any doses of HPV vaccine or are incompletely vaccinated. Recommendation for HPV vaccine could occur during pregnancy with the administration of the vaccine postpartum. Finding a way to make it easy for women to present for vaccination is imperative as this is currently a 3-vaccine series. The investigators are interested in understanding if women would find it acceptable if the investigators discussed and encouraged the vaccine while pregnant with receipt of the vaccine through their child's pediatrician at well-child visits in the postpartum period. The investigators will survey women in the third trimester of pregnancy to determine if they would find this acceptable and follow-up with them after their child's two month pediatric visit to reevaluate their opinion. No doses of the vaccine will be given.

The investigators are also interested in understanding other factors that could affect whether or not women would be interested in receiving the HPV vaccine postpartum. This includes rates of attendance at postpartum visits as well as behavioral, knowledge and demographic characteristics that may be associated with acceptability of receiving the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 28 weeks of gestational age or greater

Exclusion Criteria:

* Primary language other than English or Spanish
* Receipt of any prior doses of HPV vaccine.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women will be recruited from the hospital based UNC Obstetric and Gynecology (UOG) Clinic including the resident clinic, faculty clinics and maternal fetal medicine clinics. The UOG Clinic cares for a diverse population of women from the immediate geographical area as well as referrals from 14 surrounding funded health centers.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Acceptability of HPV vaccination | At time of enrollment
  Estimation of the proportion of women indicating that they would be willing to receive the HPV vaccine postpartum at pediatric well-child visits if offered in the third trimester of pregnancy

SECONDARY OUTCOMES:
Proportion of women attending postpartum visits | At time of follow-up which will occur 8 weeks after delivery. This could occur up to 5 months after enrollment.
  Estimation of the proportion of women who attend postpartum visits with their obstetric care providers
Estimate of baseline prevalence of prior HPV vaccination in study population | at time of enrollment
  Participants eligible for participation based on maternal age and gestational age will be screened for prior doses of HPV vaccine by self-report. Number of participants with self-report of prior HPV vaccination will be recorded and baseline prevalence from our population will be determined.

OTHER OUTCOMES:
Attitudes and beliefs regarding HPV immunization | at time of enrollment
  This will be assessed using the Carolina HPV Immunization Attitudes and Belief Scale
Health Literacy | at time of enrollment
  Health literacy will be screened using the "Newest Vital Sign" Measure
HPV and HPV vaccine Knowledge | at time of enrollment
  A series of questions will be used to determine baseline knowledge of HPV and HPV vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kilfoyle, MD, Principal Investigator — University of North Carolina, Chapel Hill; Lisa Rahandale, MD, Study Chair — University of North Carolina, Chapel Hill